CLINICAL TRIAL: NCT06656689
Title: Prospective Observational Study on Water Vapor Thermal Therapy in Management of Patients with Benign Prostatic Hyperplasia (BPH)
Brief Title: Study on Water Vapor Thermal Therapy
Status: Recruiting | Type: Observational
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Hee Youn Kim, Associate Professor, Saint Vincent's Hospital, Korea
Other Study IDs: SVHWVTT
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Rezum; Water Vapor Thermal Therapy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rezum Group: Patients who underwent Rezum water vapor thermal therapy treatment for BPH
  Interventions: Procedure: Rezum (water vapor thermal therapy)

INTERVENTIONS:
Procedure: Rezum (water vapor thermal therapy) — Rezum or water vapor thermal therapy is a procedure that involves injecting steam at 103°C into the prostate tissue to induce necrosis and reduce the size of the enlarged prostate.

SUMMARY:
The goal of this observational study is to learn about the efficacy of Rezum water vapor thermal therapy in benign prostatic hyperplasia patients. The main question it aims to answer is:

* Is Rezum an effective treatment?
* Is Rezum safe?

Participants will be followed up for at least three months after the treatment to evaluate efficacy and safety.

DETAILED DESCRIPTION:
This prospective cohort study aims to evaluate the safety and efficacy of the Rezum procedure, a minimally invasive treatment for benign prostatic hyperplasia (BPH) that utilizes convective water vapor thermal energy. The Rezum procedure was approved by the U.S. FDA in 2015, and recent approval by South Korea's Ministry of Health and Welfare has allowed its use in South Korean patients. Unlike other BPH treatments, Rezum delivers steam at 103°C directly into the prostatic tissue, inducing necrosis and reduction of prostate size through a controlled thermal effect. This process is conducted in a day-surgery setting under local, general, or spinal anesthesia, minimizing patient burden and recovery time.

The study will enroll male patients aged 50 or older with confirmed BPH who meet specific prostate size criteria, measured via transrectal ultrasound. Following a preoperative evaluation, including prostate size, PSA levels, symptom questionnaires, and urodynamic assessment, patients will undergo the Rezum procedure. This involves cystoscope-guided needle insertion into hypertrophic prostate regions, where targeted thermal energy is delivered in short bursts. The procedure is completed within a single hospital visit, and patients are generally discharged on the same day unless complications arise.

After surgery, participants will have routine follow-up visits, including catheter removal and initial voiding assessments within one week. Further follow-up, at a minimum of three months, will include standardized assessments of voiding function, symptom severity (IPSS, IIEF, OAB-q), prostate size, uroflowmetry, and residual urine volume. The safety profile will be assessed by recording adverse events, including infection, hematuria, voiding dysfunction, and the necessity for catheter reinsertion. Complications will be classified according to the Clavien-Dindo classification system.

Data analysis will assess the preoperative and postoperative changes in symptom severity, functional parameters, and prostate measurements. Comparisons of these continuous variables will utilize paired sample t-tests or Wilcoxon signed-rank tests, depending on normality test results. Variables include IPSS, IIEF, OAB-q, prostate size, PSA, maximum flow rate (Qmax), and post-void residual volume (PVR). Additionally, multiple regression analysis will identify factors contributing to the need for postoperative catheter reinsertion. Statistical significance will be set at α=0.05, with p-values below 0.05 indicating significant differences.

This study will address a current gap in research on the Rezum procedure's impact on Korean patients, contributing to the understanding of this minimally invasive approach within different populations and expanding its potential applicability.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Prostate size between 30cc and 80cc as measured by transrectal ultrasound
* Patients scheduled for Rezum surgery for BPH

Exclusion Criteria:

* Suspected prostate cancer
* Suspected urinary tract infection
* Inability to complete follow-up
* Patients who do not consent to participate in the study

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects are patients requiring surgery for benign prostatic hyperplasia (BPH).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | From enrollment to three months after treatment
  International Prostate Symptom Score (IPSS) is a validated, reproducible scoring system to assess disease severity and response to therapy for BPH. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Qmax | From enrollment to three months after treatment
  Maximal urine flow rate in uroflowmetry exam

SECONDARY OUTCOMES:
Complications | Three months after treatment
  Complications evaluated using the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Hee Youn Kim, M.D., Ph.D., Principal Investigator — St Vincent's Hospital
Locations (1):
- Saint Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request to the PI. The investigators do not have a specific URL to provide the information.

REFERENCES:
- [Background] McVary KT, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Pliskin M, Beahrs JR, Prall D, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Tadros NN, Gange SN, Roehrborn CG. Final 5-Year Outcomes of the Multicenter Randomized Sham-Controlled Trial of a Water Vapor Thermal Therapy for Treatment of Moderate to Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2021 Sep;206(3):715-724. doi: 10.1097/JU.0000000000001778. Epub 2021 Apr 19. PMID 33872051